CLINICAL TRIAL: NCT06406049
Title: FINISHING HIV: an Ending the HIV Epidemic (EHE) Model for Latinx Integrating One-Stop-Shop Pre-Exposure Prophylaxis (PrEP) Services, a Social Network Support Program and a National Pharmacy Chain
Brief Title: Finishing HIV Project
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Mariano Juan Kanamori Nishimura, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20220377; R01AI169643 (NIH)
Record Dates: First submitted 2024-05-02; First posted 2024-05-09 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-05

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- I want "Yo Quiero" Control Group (Active Comparator): Participants will receive the standard of care for up to 15-months
  Interventions: Other: Control group
- Friend "Amigx" Social network intervention (Experimental): Participant will receive a social network intervention for up to 15-months
  Interventions: Behavioral: Social network intervention

INTERVENTIONS:
Other: Control group — Participants will receive the standard of care (beginning of the study) which includes sexual health information once in-person for up to 15 minutes for the duration of the study.
  Arms: I want "Yo Quiero" Control Group
Behavioral: Social network intervention — Participants will come to the study location for up to 2 hours three times (beginning of the study, 6-month and 12-month follow-ups) during the duration of the study. During the study, participants will receive sexual health counseling for HIV prevention. Additionally participants will receive information and resources for PrEP usage. Participants will be encouraged to share sexual health information two times (three and nine months after the beginning of the study) during the duration of the study.
  Arms: Friend "Amigx" Social network intervention

SUMMARY:
This study aims to learn how to help enable healthy behaviors and lower the risk of HIV among Latinx Men.

ELIGIBILITY:
Inclusion Criteria

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Being 18 to 54 years of age
4. Being a cis-gender male
5. Self-report one or more of the following behaviors and health conditions in the last 6 months which meet the Centers for Disease Control and Prevention (CDC) clinical guidelines for PrEP eligibility

   * Diagnosed with bacterial sexually transmitted infection (e.g., syphilis, gonorrhea, or chlamydia)
   * Sex with a partner who is living with HIV
   * Sex without a condom with two or more partners whose HIV status were unknown
   * Injection drug use and sharing injection equipment
6. Self-reported status as HIV negative
7. Willing to be tested for HIV

Exclusion Criteria

1. Display diminished capacity to consent because of:

   * An inability to provide informed consent (e.g., cognitive impairment)
   * Severe psychiatric symptoms (e.g., mania, psychosis) that impair capacity to provide informed consent, as assessed by interviewers with Collaborative Institutional Training Initiative (CITI) Human Subjects Research and National Institutes of Health (NIH) Good Clinical Practice training
2. <18 years old or >54 years old
3. Self-reported living with HIV
4. Reactive HIV test (for "Amigx" seeds or "Yo Quiero" control participants)
5. Refusal of HIV test
6. Identifies as Non-Latinx
7. Individuals enrolled in other PrEP initiation interventions
8. Individuals with an active PrEP prescription in the last 6-months (oral or injectable)

Ages: 18 Years to 54 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 624 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2029-11-15 (Estimated); Study Completion 2029-11-15 (Estimated)

PRIMARY OUTCOMES:
Number of participants that report using PrEP | Up to 12-months
  PrEP initiation will be measured by analyzing the number of participants that initiate PrEP divided by the total number of participants
Number of Dried Blood Spot (DBS) tests that report PrEP use | Up to 12-months
  PrEP initiation will be measured by analyzing the number of DBS tests that report PrEP use divided by the total number of participants
Number of participants that bring a proof of PrEP prescription | Up to 12-months
  PrEP initiation will be measured by analyzing the number of participants that bring proof of a PrEP prescription divided by the total number of participants

SECONDARY OUTCOMES:
PrEP knowledge measured by PrEP knowledge question | Up to 12-months
  Scores range from 1 (I don't know) to 5 (99% or more than 99% effective). Higher scores indicate adequate PrEP knowledge.
Number of Dried Blood Spot (DBS) tests that report adequate PrEP adherence | Up to 12-months
  PrEP adherence will be measured by analyzing the number of DBS tests that report PrEP adherence divided by the total number of participants that initiate PrEP during the study

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Kanamori, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No